CLINICAL TRIAL: NCT03147508
Title: Investigating Clinical Indicators of Spine Related Dysfunction Patterns. A Clinical Study on Neck Pain Patients.
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/0971
Record Dates: First submitted 2016-09-22; First posted 2017-05-10 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Neck Pain; Neck Disorders
Keywords: Diagnostics, clinical criteria, clincal reasoning, neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week

GROUPS / COHORTS (1):
- Neck pain patients

SUMMARY:
The goal of is this study is to investigate the reliability and validity of a classification system for neck pain patients. In a previous study clinical experts were asked about the clinical criteria they considered to be determinative for 5 predefined dysfunction patterns in patients with neck problems: 1) articular, 2) myofascial, 3) neural, 4) central, and 5) sensorimotor control dysfunction pattern. This Delphi survey revealed a list of pertinent anamnestic and clinical criteria per dysfunction pattern.

In the present study we will collect anamnestic and clinical data of 200 neck pain patients. This will be obtained by approximately 20 clinicians that fill out a standardized registration form at the intake of their patients with neck pain.

The therapists and patients will receive an informed consent that clarifies the purpose of the study and what happens next with the collected data.

Per patient the therapist indicates the dominant clinical pattern based on his/her experience. Prior to the data analysis, the researchers will be blinded to the patient identification data. Subsequent, the registration forms will be screened for the presence of clinical criteria (obtained from previous Delphi study), independent of the therapist's diagnosis/conclusions. A second independent researcher will gather this information, which will be used for statistical analysis, in order to investigate which clinical criteria can be considered as determinative for a particular pattern. Outcome measures for these analysis are:

* sensitivity and classification specificity
* (positive and negative) likelihood ratios
* odds ratios
* diagnostic accuracy

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from neck pain

Exclusion Criteria:

Known serious underlying pathology (RED FLAGS):

cancer, metastatsis, untreated fractures, history of diabetes or pathology of the central nervous system, non-musculoskeletal neck pain

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from neck pain
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2016-09; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Anamnestic criteria_administrative data (descriptive) | 1 single time at first intake
  i.e. name of the patient, date of birth, sex, BMI, profession, hobbies
anamnestic criteria_ red flag screening (descriptive) | 1 single time at first intake
  i.e. a list of signs and symptoms that could refer to a severe underlying pathology
anamnestic criteria_ body chart (descriptive) | 1 single time at first intake
  i.e. a body map where pain localization, referred pain areas and the quality of the pain are registered
anamnestic criteria_ movement restriction(s) (descriptive) | 1 single time at first intake
  i.e. all movements that are limited due to the patients neck complaints are registered
anamnestic criteria_ onset and evolution of the neck complaints (descriptive) | 1 single time at first intake
  i.e. the onset and the evolution of the neck complaints are registered
anamnestic criteria_ better/worse section (descriptive) | 1 single time at first intake
  i.e. all activities that provoke and/or reduce the neck complaints are listed
anamnestic criteria_ history (descriptive) | 1 single time at first intake
  i.e. the previous episodes of similar complaints are registered
anamnestic criteria_ previous treatment (descriptive) | 1 single time at first intake
  i.e. previous treatments for similar complaints are recorded
anamnestic criteria_ yellow flags (descriptive) | 1 single time at first intake
  i.e. beliefs and appraisals of the patient which may lead to chronic neck pain are registered
anamnestic criteria_ results of additional (technical) investigations (descriptive) | 1 single time at first intake
  i.e. results of medical imagery, EMG testing, blood test that are available to the patient are collected
clinical examination criteria_ inspection & palpation (descriptive) | 1 single time at first intake
  i.e. inspection of the overall posture of the head and neck, and palpation of the soft tissues in that area to appreciate the muscle tone, temperature, swelling
clinical examination criteria_ basic functional assessment of the neck and shoulder (descriptive) | 1 single time at first intake
  i.e. active and passive movement examination of the neck and shoulder to assess the range of motion, pain, and quality of movement
clinical examination criteria_ additional testing for articular involvement (descriptive) | 1 single time at first intake
  i.e. passive intervertebral provocation and movement testing of the spinal segments of the neck
clinical examination criteria_ additional testing for myofascial involvement (descriptive) | 1 single time at first intake
  i.e. assessment of the muscle length, strength, pain provocation in tender points
clinical examination criteria_ additional testing for neurological involvement (descriptive) | 1 single time at first intake
  i.e. neurodynamic testing: palpation of the peripheral nerves in the upper limb, upper limb tension tests, reflex testing, motor and sensory function
clinical examination criteria_ additional testing for central involvement (descriptive) | 1 single time at first intake
  i.e. the NDI and CSI questionnaire
clinical examination criteria_ sensory motor control involvement (descriptive) | 1 single time at first intake
  i.e. examination of the neuromuscular control of the cervical flexor and extensor muscles
clinical examination criteria_ additional testing for other areas related to the patient's neck complaints (descriptive) | 1 single time at first intake
  i.e. temporomandibular joint / thoracic spine / lumbar spine / lower limb / abdominal examination
Clinical reasoning variables_ tissue mechanisms (descriptive) | 1 single time at first intake
  i.e. the interpretation of the therapist on the dominant tissue mechanism (nociceptive - mechanical - neuropathic - central pain) is registered
Clinical reasoning variables_ pain mechanisms (descriptive) | 1 single time at first intake
  i.e. the interpretation of the therapist on the dominant pain mechanism (input-processing-output) for that particular patient is registered, as described in a study by Gifford et al., 1998; Butler, 2000
Clinical reasoning variables_ dominant dysfunction pattern (descriptive) | 1 single time at first intake
  i.e. the presence of a cluster of findings that raise suspicion of a dominant dysfunction pattern as described in a previous study by Dewitte et al., 2016

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dewitte V, Peersman W, Danneels L, Bouche K, Roets A, Cagnie B. Subjective and clinical assessment criteria suggestive for five clinical patterns discernible in nonspecific neck pain patients. A Delphi-survey of clinical experts. Man Ther. 2016 Dec;26:87-96. doi: 10.1016/j.math.2016.07.005. Epub 2016 Jul 21. PMID 27507590
- [Derived] Dewitte V, De Pauw R, Danneels L, Bouche K, Roets A, Cagnie B. The interrater reliability of a pain mechanisms-based classification for patients with nonspecific neck pain. Braz J Phys Ther. 2019 Sep-Oct;23(5):437-447. doi: 10.1016/j.bjpt.2018.10.008. Epub 2018 Oct 29. PMID 30389348